CLINICAL TRIAL: NCT06354803
Title: Amelioration of Kinaesthesia in Pregnant Women Using Pezzi Ball Exercises: Randomized Controlled Trial
Brief Title: Effect of Pezzi Ball on Balance in Pregnant Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed elsaied moghazy ahmed, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KafrelsheikhU 30
Record Dates: First submitted 2024-03-12; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Postural Stability
Keywords: Kinaesthetic training

STUDY DESIGN:
Intervention Model Description: 45 participants with gestational age below 28 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drawing procedure was conducted by a researcher without disclosure to the participants, ensuring unbiased allocation. Moreover, both the assessor and statistician remained blinded throughout the assessment period, unaware of the group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): 23 women below 28 week gestation were received kinaesthetic exercises on the Pezzi ball and standard antenatal care
  Interventions: Other: proprioceptive training
- control group (No Intervention): 22 women belowe 28 week gestation were received just standard antenatal care

INTERVENTIONS:
Other: proprioceptive training — Proprioceptive training using swiss ball for 12 sessions
  Other Names: Standard antenatal care
  Arms: intervention group

SUMMARY:
The effect of kinaesthetic training on performance and postural stability during pregnancy and 2 weeks postpartum

DETAILED DESCRIPTION:
The effect of kinaesthetic training using pezzi ball for 12 sessions with rate of 3 session per week on postural stability and performance during pregnancy and at the 2-week postpartum follow-up. Postural stability was measured using a balance check board 636-1

ELIGIBILITY:
Inclusion Criteria:

* age between 25 and 30 years a body mass index (BMI) not exceeding 32 kg/m2, low-risk gestation primiparous pregnancy intact sensory motor integration in the lower extremities.

Exclusion Criteria:

* more than 28 weeks gestation
* had chronic disease
* multiparous

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnanc women
Enrollment: 45 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
change of postural stability | 1 month
  By the use of balance check board 636-1 the balance of pregnant women changed significantly which appears in change in the rate of falling

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy kafrelshiekh university, Kafr ash Shaykh, Kafrelshiekh, Egypt